CLINICAL TRIAL: NCT05307341
Title: Improving Pain Management and Decreasing Length of Stay After THA and TKA: A Randomized, Patient-Blinded Comparison of Standard of Care Pain Management With and Without Sufentanil
Brief Title: Improving Pain Management and Decreasing LOS After Total Hip Arthroplasty (THA) and Total Knee Arthroplasty (TKA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: More Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain20210928.3
Record Dates: First submitted 2022-01-27; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: pain; length of stay; peri-operative; THA; TKA
MeSH Terms: conditions — Pain | interventions — Sufentanil; Dsuvia

STUDY DESIGN:
Intervention Model Description: two arm, patient blinded, randomized, post market
Who Masked: Participant
Masking Description: participant will not be informed whether participant is in the standard of care arm or treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): One dose of sufentanil 30 mcg sublingual will be given pre-operatively when entering the operating room and one dose post-operatively in the PACU in addition to standard of care pain management.
  Interventions: Drug: sufentanil
- Control (No Intervention): A multimodal approach to analgesia will be used in all subjects in the perioperative setting and will be used in both the control and treatment groups. Intraoperative dosing of opioids will be based on the anesthesiologist's clinical judgement related to the pain and hemodynamic response to surgical stimuli and on an as needed basis in the PACU. Administration of opioids in the PACU will be in response to moderate-to-severe pain.

INTERVENTIONS:
Drug: sufentanil — One dose of sufentanil 30 mcg sublingual pre-operatively upon entry to operating room and one dose of sufentanil 30 mcg sublingual in the PACU.
  Other Names: sufentanil (DSUVIA)
  Arms: Treatment

SUMMARY:
This two arm, patient blinded, randomized, post market clinical trial in a single orthopedic hospital will determine whether there is improved pain management and decreased length of stay when comparing standard of care pain management with and without sufentanil.

DETAILED DESCRIPTION:
This two arm, patient blinded, randomized, post market clinical trial in a single orthopedic hospital will determine whether there is improved pain management and decreased length of stay (LOS) when comparing standard of care pain management with and without sufentanil. The objective is to compare LOS between patients who have had primary THA or TKA and have received standard of care peri-operative pain management and one dose of sufentanil 30 mcg sublingual pre-operatively in the operating room and one dose post-operatively in the post anesthesia care unit (PACU) versus those who have received only standard of care peri-operative pain management in a orthopedic specialty hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 50 to 80 years, inclusive
2. Planned primary THA or TKA
3. Expressed willingness to be discharged the same day of surgery if condition allows
4. American Society of Anesthesiologists (ASA) physical classes I - III

   1. ASA I: A normal healthy patient. Example: Fit, nonobese (BMI under 30), a nonsmoking patient with good exercise tolerance.
   2. ASA II: A patient with a mild systemic disease. Example: Patient with no functional limitations and a well-controlled disease (e.g., treated hypertension, obesity with BMI under 35, frequent social drinker or is a cigarette smoker).
   3. ASA III: A patient with a severe systemic disease that is not life-threatening. Example: Patient with some functional limitation as a result of disease (e.g., poorly treated hypertension or diabetes, morbid obesity, chronic renal failure, a bronchospastic disease with intermittent exacerbation, stable angina, implanted pacemaker).
5. Patients who are English competent.

Exclusion Criteria:

1. Opioid tolerant (> 50 mg oral morphine milligram equivalents (MMEs) daily)
2. Current IV drug abuse
3. History of alcoholism
4. History of severe renal impairment
5. History of severe hepatic impairment
6. Dependent on supplemental oxygen at home
7. Pregnant
8. Incarcerated
9. Patient unable to provide informed consent
10. Patients undergoing bilateral TKA, THA
11. Patient undergoing unicompartmental knee arthroplasty (UKA)
12. Patients undergoing other concurrent surgery
13. Patients with a history of allergy to any drugs in the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Length of stay | From date and time of hospital admission until date and time of hospital discharge, assessed up to 3 days after hospital admission
  length of hospital stay
Discharge location | At date of discharge from hospital, assessed up to 3 days after hospital admission
  Discharged from the PACU instead of the Medical-Surgical Unit

SECONDARY OUTCOMES:
morphine milligram equivalent (MME) doses | From date and time of hospital admission until date and time of hospital discharge, assessed up to 3 days after hospital admission
  the amount of MME doses received
side effect(s) | From date and time of hospital admission until date and time of hospital discharge, assessed up to 3 days after hospital admission
  opioid related side effects
physical therapy | From admission date and time in PACU until discharge date and time from PACU, assessed for 12 hours after surgery
  ability to complete physical therapy in PACU
patient satisfaction | At date and time of discharge from the hospital, within 3 days following hospital admission
  patient reported satisfaction of pain management on a 4-point Likert scale with a higher score being more satisfied
hospital costs | From date of hospital admission until date of hospital discharge, assessed for 3 days following hospital admission
  total hospital costs

CONTACTS AND LOCATIONS:
Overall Officials: Debra Sietsema, PhD, Study Director — More Foundation
Locations (1):
- The CORE Institute Specialty Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No